CLINICAL TRIAL: NCT04661163
Title: The CHALLENGE-trial: the Effects of a Virtual Reality-assisted Exposure Therapy for Persistent Auditory Hallucinations Versus Supportive Counselling in People With Psychosis
Brief Title: CHALLENGE. A Randomised Clinical Trial Examining Virtual Reality Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Region of Southern Denmark (Other); Mental Health Services in the North Denmark Region (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHALLENGE
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Auditory Hallucinations
Keywords: Avatar; Schizophrenia; Auditory Hallucinations; Psychotherapy; Virtual Reality; Psychosis; Virtual Reality Therapy
MeSH Terms: conditions — Hallucinations; Schizophrenia; Psychotic Disorders | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: A randomised, assessor-blinded parallel-groups superiority clinical trial
Who Masked: Outcomes Assessor
Masking Description: Independent assessors blinded to the treatment will evaluate outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality avatar therapy (Experimental): Patients will be offered seven individual sessions of virtual reality therapy and two booster sessions conducted by a skilled therapist. In the initial phase of treatment, the participants create a virtual avatar that corresponds to their visual perception of the source of their voice. The therapist initiates, encourages and supports a dialogue between the participant and the avatar by alternating between talking as the avatar and as a supportive therapist. The therapy sessions last 50 minutes of which around 15 minutes is spent in dialogue with the avatar. The remaining 30 minutes will be used on preparing the patient for the confrontation with the avatar, evaluating on the interaction with the avatar, and use general cognitive behavioral techniques to reduce the auditory hallucination. The treatment is conducted with the use of virtual reality, so the participant will wear VR headset during treatment and watch and talk with the avatar shown in front of him or her.
  Interventions: Other: Psychotherapy
- Supportive counselling (comparison group) (No Intervention): The control group is offered seven session with health professionals providing supportive counselling. This can (but does not necessarily) involve psychotherapy targeting auditory hallucinations.

INTERVENTIONS:
Other: Psychotherapy — Virtual Reality Avatar Therapy is a psychotherapeutic intervention targeting auditory hallucinations
  Other Names: Virtual Reality Avatar Therapy
  Arms: Virtual reality avatar therapy

SUMMARY:
The study is a randomised, assessor-blinded parallel-groups superiority clinical trial, allocating a total of 266 patients to either the experimental intervention or standard intervention. The participants will be randomised to either 12-weeks of virtual reality therapy or supportive counselling. All participants will be assessed at 12- and 24 weeks post baseline. A stratified block-randomisation with concealed randomisation sequence will be conducted. Independent assessors blinded to the treatment will evaluate outcome. Analysis of outcome will be carried out with the intention to treat principles.

DETAILED DESCRIPTION:
Auditory hallucinations are among the most frequent symptoms in psychotic disorders. While a large group of patients with first episode psychosis achieve remission of psychotic symptoms during first year after initial contact with mental health services, almost one third continue having psychotic symptoms in spite of treatment with antipsychotic medication. Since auditory hallucinations are a major cause of distress and suffering for these patients, there is an essential need to test the effectives of targeted psychotherapeutic interventions in alleviating auditory hallucinations Two previous trials have provided preliminary evidence of the effectiveness of virtual reality therapy on auditory hallucinations, but no trial to date has examined the effect of virtual reality assisted therapy in an adequately powered RCT. In this large-scale randomized, clinical trial, patients in the experimental intervention will be receiving 7 sessions of virtual reality assisted avatar therapy while patients in the control group will receive 7 sessions of supportive contact with mental health care professionals at their regular outpatient clinic.

If the virtual reality therapy is found to be beneficial in reducing the severity of refractory auditory hallucinations, it will be a breakthrough in the current treatment of psychotic disorders. A large group of patients with schizophrenia and related disorders in Denmark and worldwide will be the target group of the therapy. If proven effective, the treatment will be especially relevant for patients with treatment resistant schizophrenia, but the treatment can also be used as an add on to antipsychotic medication for patients with a better prognosis, such as patients with first episode psychosis. If the virtual reality therapy is proven effective, it can be implemented in mental health services in Denmark and internationally. A successful implementation could reduce the costs associated with treatment of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - years
2. Ability to give informed consent
3. A schizophrenia spectrum disorder (ICD-10 code: F20 -F29)
4. Auditory hallucinations for at least three months, corresponding to a SAPS score on auditory hallucinations of ≥3.
5. No changes in antipsychotic medication within the past four weeks and

   1. Not responding to current antipsychotic compound or
   2. Not responding to at least two antipsychotic compounds. Table2

Exclusion Criteria:

1. Rejecting informed consent
2. Unable to identify a single dominant voice to work on
3. A diagnosis of organic brain disease
4. Substance to a level that hinders engagement in therapy.
5. Auditory hallucinations in a language not spoken by the therapists
6. A command of spoken Danish or English inadequate for engaging in therapy
7. Inability to tolerate the assessment process
8. Strongly impaired vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Level of auditory hallucinations | 12 weeks from inclusion
  Level of auditory hallucinations measured with The Psychotic Symptoms Rating Scales (PSYRATS-AH) total score at cessation of treatment at 12-weeks (score on PSYRATS-AH: 0-44. A score of 0 is the minimum score and 44 is the maximum score i.e. a score of 44 is the worst possible outcome.

SECONDARY OUTCOMES:
Frequency of auditory hallucinations | 12 weeks from inclusion
  PSYRATS-AH-Frequency.
Distress caused by auditory hallucinations | 12 weeks from inclusion
  PSYRATS-AH-Distress
Voice acceptance | 12 weeks from inclusion
  Questionnaire: the Voices Acceptance and Action Scale (VAAS-Action)
Assertive Responding to Voices | 12 weeks from inclusion
  Questionnaire: Assertive Responding to Voices (Approve - Voices), The assertive subscale (5 items with scores from 0-10, minimum score on this subscale is 0, maximum score is 50 with higher scores being a better outcome)
Personal and social performance | 12 weeks from inclusion
  The personal and social performance scale (PSP); (Scores from 1-100, with a score of 100 being the best possible outcome).
Perceived voice power | 12 weeks from inclusion
  Questionnaire: Voice Power Differential Scale, total score (range 7-35 with 7 being the minimum score and 35 the maximum score. Higher scores indicates greater power differential in favour of the voice - i.e. a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, professor, Principal Investigator — Mental Health Services Capitol of Denmark; Copenhagen Research Center for Mental Health - CORE
Locations (1):
- Copenhagen Research Center for Mental Health - CORE, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith LC, Vernal DL, Mariegaard LS, Christensen AG, Jansen JE, Schytte G, Stokbro LA, Albert N, Christensen MJ, Thomas N, Hjorthoj C, Nordentoft M, Glenthoj LB. Immersive virtual reality-assisted therapy targeting persistent auditory verbal hallucinations in patients diagnosed with schizophrenia spectrum disorders in Denmark: the Challenge assessor-masked, randomised clinical trial. Lancet Psychiatry. 2025 Aug;12(8):557-567. doi: 10.1016/S2215-0366(25)00161-0. Epub 2025 Jul 3. PMID 40617245